CLINICAL TRIAL: NCT05273645
Title: World-wide Survey on the Incidence, Diagnosis and Prognosis of Atrio-oesophageal Fistula Following Percutaneous Catheter Ablation
Brief Title: PrOgnosis Following Esophageal FisTula FormaTion in Pts Undergoing CathetER Ablation for AF Study
Acronym: POTTER
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Roland Richard Tilz, MD, Prof. Dr. med. Roland Richard Tilz, University of Luebeck
Other Study IDs: Potter AF Study
Record Dates: First submitted 2022-02-21; First posted 2022-03-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Atrio-Oesophageal Fistula; PVI; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Pulmonary vein isolation emerged as an effective and safe strategy to treat atrial fibrillation patients. Atrio-oesophageal fistula (AOF) represents a rare but devastating complication of AF ablation procedure. This complication (0.016-0.07%) requires an international effort to allow for better understanding of the factors contributing to its occurrence and the best management strategies. A worldwide, retrospective, multicenter registry focusing on the incidence, diagnosis and management of this complication.

DETAILED DESCRIPTION:
Data about the incidence, optimal management and outcome of AOF is sparse. The largest national and international surveys report on less than 50 AOF. The latest worldwide survey was conducted in 2015 and managed to include 31 patients who developed AOF after atrial fibrillation ablation procedure. In the meanwhile, the total number of AF ablation procedures increased significantly. Additionally, AF ablation technology changes significantly with e.g. increasing numbers of cryoballoon ablation and contact force guided radiofrequency ablation.

The study is designed as a worldwide, multi-centre, anonymised registry study to evaluate the incidence, optimal management and outcome of this AOF. More than 50 patients with AOF following percutaneous catheter ablation will be included in the register.

ELIGIBILITY:
Inclusion Criteria:

* Atrio-oesophageal fistula after Ablation
* Indication for AF ablation as per current guidelines
* Performing the ablation at an ablation centre

Exclusion Criteria:

* No Atrio-oesophageal fistula after Ablation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing PVI and developing an AOF
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence of AOF following percutaneous catheter ablation | 5 year
  1. Evaluating the Incidence of atrio-oesophageal fistula after percutaneous catheter ablation in patients with atrial fibrillation, as well as the more detailed analysis of the incidence of AOF after PVI with Cryo Balloon or RF Contact Force

SECONDARY OUTCOMES:
Diagnosis and management of AOF | 5 year
  Evaluating the diagnosis and management of the AOF
Mortality rate | 5 year
  Analysis of the mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Tilz, Principal Investigator — Universitaet Luebeck
Locations (1):
- Klinik für Rhythmologie, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tilz RR, Schmidt V, Purerfellner H, Maury P, Chun KRJU, Martinek M, Sohns C, Schmidt B, Mandel F, Gandjbakhch E, Laredo M, Gunawardene MA, Willems S, Beiert T, Borlich M, Iden L, Futing A, Spittler R, Gaspar T, Richter S, Schade A, Kuniss M, Neumann T, Francke A, Wunderlich C, Shin DI, Meininghaus DG, Foresti M, Bonsels M, Reek D, Wiegand U, Bauer A, Metzner A, Eckardt L, Popescu SS, Krahnefeld O, Sticherling C, Kuhne M, Nguyen DQ, Roten L, Saguner AM, Linz D, van der Voort P, Mulder BA, Vijgen J, Almorad A, Guenancia C, Fauchier L, Boveda S, Greef Y, Da Costa A, Jais P, Derval N, Milhem A, Jesel L, Garcia R, Poty H, Khoueiry Z, Seitz J, Laborderie J, Mechulan A, Brigadeau F, Zhao A, Saludas Y, Piot O, Ahluwalia N, Martin C, Chen J, Antolic B, Leventopoulos G, Ozcan EE, Yorgun H, Cay S, Yalin K, Botros MS, Mahmoud AT, Jedrzejczyk-Patej E, Inaba O, Okumura K, Ejima K, Khakpour H, Boyle N, Catanzaro JN, Reddy V, Mohanty S, Natale A, Blessberger H, Yang B, Stevens I, Sommer P, Veltmann C, Steven D, Vogler J, Kuck KH, Merino JL, Keelani A, Heeger CH. A worldwide survey on incidence, management, and prognosis of oesophageal fistula formation following atrial fibrillation catheter ablation: the POTTER-AF study. Eur Heart J. 2023 Jul 14;44(27):2458-2469. doi: 10.1093/eurheartj/ehad250. PMID 37062040